CLINICAL TRIAL: NCT05834426
Title: Omic Technologies Applied to the Study of Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma for the Discovery of Diagnostic and Prognosis Biomarkers
Brief Title: Omic Technologies Applied to the Study of B-cell Lymphoma for the Discovery of Diagnostic and Prognosis Biomarkers
Status: Not yet recruiting | Type: Observational
Sponsor: Sociedad de Lucha Contra el Cáncer del Ecuador (Other)
Responsible Party: Sponsor
Other Study IDs: CISOLGYE20230021
Record Dates: First submitted 2023-04-03; First posted 2023-04-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, B-Cell; Neoplasms; Cancer; High-grade B-cell Lymphoma; Diffuse Large B Cell Lymphoma; Non Hodgkin Lymphoma; Metabolomics
Keywords: Metabolomic Analysis
MeSH Terms: conditions — Lymphoma, B-Cell; Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples from patients with Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma at diagnosis, during and after treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Plasma metabolomic profile by Ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry (UPLC-QTOFMS) — For metabolomic analysis, different portions of the blood (plasma and lymphocytes) will be subjected to metabolite extraction by the extraction method defined by Glasgow Polyomics. With protein precipitation, 200 microliters (uL) of the fluid with the metabolites is transferred to a new microtube and must be maintained at -80 °C until the time of metabolomic analysis.

SUMMARY:
The goal of this observational study is to determine the plasma metabolomic profile in diffuse large B-cell lymphoma and high-grade B lymphomas patients before, during and after treatment by ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry (UPLC-QTOFMS)

DETAILED DESCRIPTION:
The main question it aims to answer is the correlation between the plasma metabolomic profile of diffuse large B-cell lymphoma and high-grade B lymphomas patients before and after treatment determined by ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry (UPLC-QTOFMS) and analysed with MetaboAnalyst web platform to identify specific over- or under-expressed markers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older;
* Both sexes;
* Patients with confirmed histopathological diagnosis of Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2;
* Patient intending to receive full-dose treatment (Monoclonal antibodies plus anthracycline based combination chemotherapy);
* Staged with PET-CT or CT.

Exclusion Criteria:

* Patients with comorbidities that may interfere with the interpretation of the results (CKD in dialysis phase, Autoimmune diseases, uncontrolled Diabetes Mellitus (DM), symptomatic Heart Failure (CHF), HIV positive, positive serology for hepatitis B and C);
* Patients requiring multiple blood transfusions (4 or more blood components for the same period or cause);
* Pregnant women;
* First-line treatment in another institution;
* Diffuse transformed Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma according to the 2022 WHO classification
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma concentration as measured by ultra-high performance liquid chromatography with quadrupole time-of-flight mass spectrometry (UPLC-QTOFMS) | 12 months
  For metabolomic analysis, different portions of the blood (plasma and lymphocytes) will be subjected to metabolite extraction by the extraction method defined by Glasgow Polyomics. With protein precipitation, 200 microliters (uL) of the fluid with the metabolites is transferred to a new microtube and must be maintained at -80 °C until the time of metabolomic analysis.

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) related to the plasma metabolomic profile | 12 months
  Progression-Free-Survival calculates the time from patient treatment to disease recurrence or death due to disease progression related to the metabolomic profile during the time of observation
Prognostic factors as measured by the National Comprehensive Cancer Network International Prognostic Index (NCCN-IPI) | 12 months
  The NCCN-IPI is a robust and useful tool to stratify prognostically relevant subgroups of Diffuse Large B-cell Lymphoma and High-grade B-cell Lymphoma patients in the current era of rituximab-based therapy
Correlation between change in plasma metabolomic profile and treatment response as measured by Lugano criteria by PET-CT (positron emission tomography / computer tomography) or CT (computer tomography) scan | 12 months
  A correlation between change in plasma metabolomic profile and treatment response as measured by Lugano criteria by PET-CT or CT scan will be analysed using the Pearson's and Spearman's coefficients. The Lugano classification is used for assessment, staging and response of Hodgkin lymphoma and non-Hodgkin lymphoma. Criteria responses range from complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD), with progressive disease (PD) indicating worse response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine García Matamoros, MD, Principal Investigator — Sociedad de Lucha Contra el Cáncer del Ecuador; Fernanda Bertuccez Cordeiro, PhD, Principal Investigator — Escuela Superior Politécnica del Litoral
Locations (1):
- Instituto Oncológico Nacional Dr. Juan Tanca Marengo, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian L, Li C, Sun J, Zhai Y, Wang J, Liu S, Jiang Y, Wu W, Xing D, Lv Y, Guo J, Xu H, Sun H, Li Y, Li L, Zhao Z. Efficacy of chimeric antigen receptor T cell therapy and autologous stem cell transplant in relapsed or refractory diffuse large B-cell lymphoma: A systematic review. Front Immunol. 2023 Jan 17;13:1041177. doi: 10.3389/fimmu.2022.1041177. eCollection 2022. PMID 36733398
- [Background] Nowakowski GS, Feldman T, Rimsza LM, Westin JR, Witzig TE, Zinzani PL. Integrating precision medicine through evaluation of cell of origin in treatment planning for diffuse large B-cell lymphoma. Blood Cancer J. 2019 May 16;9(6):48. doi: 10.1038/s41408-019-0208-6. PMID 31097684
- [Background] Carneiro BA, Costa R, Taxter T, Chandra S, Chae YK, Cristofanilli M, Giles FJ. Is Personalized Medicine Here? Oncology (Williston Park). 2016 Apr;30(4):293-303, 307. PMID 27085327
- [Background] Rinschen MM, Ivanisevic J, Giera M, Siuzdak G. Identification of bioactive metabolites using activity metabolomics. Nat Rev Mol Cell Biol. 2019 Jun;20(6):353-367. doi: 10.1038/s41580-019-0108-4. PMID 30814649
- [Background] Schmidt DR, Patel R, Kirsch DG, Lewis CA, Vander Heiden MG, Locasale JW. Metabolomics in cancer research and emerging applications in clinical oncology. CA Cancer J Clin. 2021 Jul;71(4):333-358. doi: 10.3322/caac.21670. Epub 2021 May 13. PMID 33982817
- [Background] Pera B, Krumsiek J, Assouline SE, Marullo R, Patel J, Phillip JM, Roman L, Mann KK, Cerchietti L. Metabolomic Profiling Reveals Cellular Reprogramming of B-Cell Lymphoma by a Lysine Deacetylase Inhibitor through the Choline Pathway. EBioMedicine. 2018 Feb;28:80-89. doi: 10.1016/j.ebiom.2018.01.014. Epub 2018 Jan 31. PMID 29396295
- [Background] Fahrmann JF, Saini NY, Chia-Chi C, Irajizad E, Strati P, Nair R, Fayad LE, Ahmed S, Lee HJ, Iyer S, Steiner R, Vykoukal J, Wu R, Dennison JB, Nastoupil L, Jain P, Wang M, Green M, Westin J, Blumenberg V, Davila M, Champlin R, Shpall EJ, Kebriaei P, Flowers CR, Jain M, Jenq R, Stein-Thoeringer CK, Subklewe M, Neelapu SS, Hanash S. A polyamine-centric, blood-based metabolite panel predictive of poor response to CAR-T cell therapy in large B cell lymphoma. Cell Rep Med. 2022 Nov 15;3(11):100720. doi: 10.1016/j.xcrm.2022.100720. PMID 36384092